CLINICAL TRIAL: NCT05202665
Title: The Evaluation of Resin Infiltration or Fluoride Varnish Effect on Non-cavited Proximal Caries Lesion Progress at Individuals Modarate/High Caries Risk
Brief Title: Resin Infiltration and Fluoride Varnish Lesion Arresting Efficacy on Non-cavitated Proximal Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, TIJEN PAMIR, Prof. Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 70198063-050.06.04/17-8/7
Record Dates: First submitted 2021-12-20; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Dental Caries on Smooth Surface Limited to Enamel; Tooth Demineralization; Dental Caries; Dentistry, Operative; Dental Caries Activity Tests; Cariogram
Keywords: Tooth Demineralization; Dental Caries; Dentistry, Operative; Dental Caries Activity Tests
MeSH Terms: conditions — Tooth Demineralization; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flouride Varnish applications (non-invasive approaches) (Experimental): ClinproTM White Varnish 22600 ppm, 3M ESPE was applied in line with the manufacturer's recommendation to non-cavitated proximal caries lesion.
  Interventions: Procedure: ClinproTM White Varnish, 3M ESPE Fluoride Varnish (non-invasive approach)
- Resin Infiltration (micro-invasive approaches) (Experimental): ICON DMG was applied in line with the manufacturer's recommendation to non-cavitated proximal caries lesion.
  Interventions: Procedure: ICON DMG Resin Infiltration (micro-invasive approach)

INTERVENTIONS:
Procedure: ICON DMG Resin Infiltration (micro-invasive approach) — A plastic wedge located below the contact point to apart from the surface from adjacent tooth. A 15% HCl etching gel (Icon, DMG, Hamburg, Germany) was applied by syringe below the contact point for 120 s. After, the gel was washed off with air-water-spray for 30 s. The lesion was desiccated by air-blowing for 10 s, application of ethanol for 30 s and air-blowing again for 30 s. A resin infiltrant (Icon, DMG, Hamburg, Germany) was applied with another plastic holder during 3 min. Following the penetration, excess of material was removed by air blowing and flossing. The resin was light-cured for 40 s total from the buccal, occlusal, and lingual/palatal aspects. It was needed to reapplicate the resin infiltration for once because of infiltrating remaining porosities during 1 minute. Excess material removing process was again repeated and light cured for 40 s.
  Arms: Resin Infiltration (micro-invasive approaches)
Procedure: ClinproTM White Varnish, 3M ESPE Fluoride Varnish (non-invasive approach) — Tooth surfaces were cleaned thoroughly and isolated with cotton rolls. According to the manufacturer's instructions, the unit dose packages were opened, and the contents were dispensed onto the application guide and mixed to avoid the separation of sodium fluoride components. A thin coat of varnish (ClinproTM White Varnish, 3M ESPE, USA) with 22600 ppm fluoride was applied to the tooth interface with a brush tip applicator and waited for 5 minutes. Aproximal areas were coated with dental floss. The patient was instructed not to rinse or apply suction immediately after application. Patients were advised to avoid eating hard and sticky foods or drinking hot beverages for the next 2 hours, to consume a soft diet immediately after 30 minutes and to avoid brushing and flossing for the rest of the day.
  Arms: Flouride Varnish applications (non-invasive approaches)

SUMMARY:
Protection of dental hard tissues is one of the most important points of cariology. For this purpose, oral hygiene training (effective brushing and motivation), non-invasive approaches such as flouride varnish applications and micro-invasive approaches such as resin infiltration technique are applied in clinical practice. In this study, the effect of resin infiltration or fluoride varnish application on lesion depth in individuals with moderate/high caries risk was investigated.

The study was a randomized controlled, prospective and parallel designed clinical trial. 60 patients were included in the study and patients were randomly allocate to the groups. Caries risk of individuals was determined according to Cariogram, which is a computer program․ According to visual clinical examination, stage the caries continuum were (ICDAS 1,2) scored and the caries diagnostic criteria scored acording to (Nyvad 1, 2, 4, 5) The teeth wich has one caries lesion in border of enamel or prolonged to first 1/3 part of dentin in bite-wing radiograph (lesion level: E1, E2, D1) included in this study. Patient's gingival condition evaluating at initial and control sessions with gingival index (0=healthy, 1=mild inflammation, 2=moderate inflammation and bleeding on pressure). Oral hygiene training was given to all subjects included in the study and the use of fluoride toothpaste (1450 ppm, NaF) was recommended. This study was performed in a single center by experienced physicians. Resin infiltration (Icon DMG, USA) was applied to one of the groups(n=30), while fluoride varnish (ClinproTM White Varnish 22600 ppm, 3M ESPE, USA) was applied to the other group(n=30). The patients follow-up time was anticipated for 60 months in 6-month periods. The inicial visual clinical examination(T0) and follow-up sessions (T 1, 2, 3, 4, 5, 6, 7, 8, 9, 10) were conducted by two experienced researchers blind to the group information. At the aim of the study, evaluation difference in non-cavited proximal lesion progression between the resin infiltration (micro-invasive) and fluoride varnish (non-invasive) treatment options at the individuals with moderate or high risk of caries.

ELIGIBILITY:
Inclusion Criteria:

* individuals with moderate/high risk of caries
* the presence of one or more noncavitated interproximal caries lesions with radiolucencies involving the outher half of enamel up to the outer third of dentin in bite-wing radiographies (lesion depth: E1, E2, D1)
* vital posterior teeth without cavitation in which the clinically active non-carious lesion had
* Only one tooth per patient was included in the study

Exclusion Criteria:

* incapable of contracting
* pregnancy
* presence of secondary caries or restoration in the involved tooth
* lack of contact teeth
* incapable of contracting

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The non-cavitated proximal caries lesion progression change as measured by radiographic lesion depth scale | The patients follow-up time was anticipated for 60 months in 6-month periods with ten intervals.
  The non-cavitated proximal carious lesion progression as measured by radiographic lesion depth scale, radiographic score change from baseline with radiographic lesion depth scale over 60 months in 6-month periods.
  Description of the radiographic lesion depth scale scores used in this study:
  E1 = radiolucency in outer half of enamel E2 = radiolucency in inner half of enamel D1= radiolucency in outer third of dentine

CONTACTS AND LOCATIONS:
Overall Officials: Elif Ercan Devrimci, PhD, Study Chair — Ege University
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Resin Infiltration of Caries Lesions — http://journals.sagepub.com/doi/10.1177/0022034510369289
- See also: MI varnish and MI paste plus in a caries prevention and remineralization study: A randomized controlled trial — http://link.springer.com/10.1007/s00784-017-2314-9